CLINICAL TRIAL: NCT03060707
Title: Comparison of Hourly Rocuronium Consumption Using Continuous Infusion Versus Intermittent Bolus Injection: a Randomized Controlled Trial
Brief Title: Continuous Infusion Versus Intermittent Bolus Injection of Rocuronium
Acronym: RCVB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Prof., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H1612-115-817
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Muscle Relaxation; Anesthesia
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous infusion (Experimental): The group of participants who are designated to receive continuously infused rocuronium.
  Interventions: Drug: Rocuronium Bromide
- Bolus administration (Active Comparator): The group of participants who are designated to receive bolus administered rocuronium.
  Interventions: Drug: Rocuronium Bromide

INTERVENTIONS:
Drug: Rocuronium Bromide — Continuously infuse, or bolus administer rocuronium.

SUMMARY:
The research is to find out whether continuous infusion of rocuronium requires more or less amount of rocuronium, per kilogram and per hour, than bolus administered rocuronium during noncardiac surgery.

DETAILED DESCRIPTION:
comparing the total dose of rocuronium between continuous infusion and intermittent injection

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged between 2 and 12, undergoing elective noncardiac surgery which requires general anesthesia but does not require intense block, and estimated time of surgery is between 2 and 5 hours

Exclusion Criteria:

* ASA class 3-6
* BMI >= 30
* Previous history of hepatic failure, renal failure or neuromuscular disease
* Patients taking medicine which interacts with rocuronium bromide, before or during surgery: aminoglycosides, lincosamides, acylamino-penicillin antibiotics, tetracyclines, metronidazole (high dose), diuretics, MAO inhibitors, calcium channel blockers, corticosteroids, phenytoin, carbamazepine, or norepinephrine
* Previous history of allergic reaction (including anaphylactic reaction) and/or malignant hyperthermia during general anesthesia
* Patients taking medicines which contains magnesium

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Rocuronium dose per kilogram per hour | end of the surgery
  Total dose of rocuronium injected during surgery, divided by patient body weight and anesthesia time.

SECONDARY OUTCOMES:
Desaturation event | Right after the patient is transferred to the ward, from PACU (1 day)
  Whether the participant's peripheral oxygen saturation (SpO2) decreased less than 93%, in postanesthesia care unit (PACU).
Surgical rating scale | end of the surgery
  Numerical scale describing how easy it is for surgeon to access surgical field, ranging from1 to 5

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi SN, Jang YE, Lee JH, Kim EH, Kim JT, Kim HS. Comparison of rocuronium requirement in children with continuous infusion versus intermittent bolus: A randomised controlled trial. Eur J Anaesthesiol. 2019 Mar;36(3):194-199. doi: 10.1097/EJA.0000000000000934. PMID 30540640